CLINICAL TRIAL: NCT02164591
Title: Escalating Temporary Gastric Electrical Stimulation for Severe Gastroparesis
Brief Title: Escalating Temporary Gastric Electrical Stimulation (GES) for Severe Gastroparesis
Acronym: TempGES
Status: Terminated | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, John M. Wo, MD, Indiana University
Other Study IDs: Temp GES
Record Dates: First submitted 2014-06-06; First posted 2014-06-16 (Estimated); Last update posted 2020-08-04 (Actual); Status verified 2020-08

CONDITIONS: Gastroparesis
Keywords: gastroparesis; gastric electrical stimulator; GES; vomiting; nausea; bloating; postprandial fullness; epigastric pain
MeSH Terms: conditions — Gastroparesis; Vomiting; Nausea

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum to be frozen
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to determine the physiologic effects of temporary gastric electrical stimulation in subjects with severe gastroparesis.

DETAILED DESCRIPTION:
This study will look to determine the clinical benefit placing temporary gastric electrical stimulation, the ability to predict the clinical response to surgical implantation of GES, and the feasibility and patient tolerability of endoscopic placement of temporary Gastric Electrical Stimulator (t-GES),

ELIGIBILITY:
Inclusion Criteria:

* At least 3 months of gastroparesis-related symptoms, such as nausea, emesis, and/or retching
* Solid phase 4-hr gastric scintigraphy is consistent with gastroparesis within 3 months of study enrollment*

  * retention at 2 hr: >60% or
  * retention at 4 hr: >10% *Based on International consensus on gastric scintigraphy

Exclusion Criteria:

* Gastric outlet, small bowel, or colon obstruction.
* Small bowel malrotation
* Inflammatory bowel disease
* Contraindication for surgical implantation of GES
* Presence of illness that may require MRI during the study; such as pituitary tumor, herniated disc, spinal stenosis, multiple sclerosis, etc.
* Significant comorbidity due to sever cardiovascular, renal, pulmonary, or liver disease.
* Significant coagulopathy
* Non-ambulatory patients: bed-ridden, nursing home resident, etc.
* Pregnancy
* Unable to give own informed consent
* Prisoners

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who have been diagnosed with gatroparesis.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2013-02; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Improvement in the symptoms of gastroparesis by t-GES in patients with severe gastroparesis. | 1 month
  Review the symptoms before and after the t-GES placements and follow for any improvement

SECONDARY OUTCOMES:
Clinical response to t-GES placement as measured by questionnaires | 1 year
  Measuring the responses to questionnaires before and after placement of GES
Develop a prospective registry in patients undergoing escalating t-GES | 1 year
  Have a database of patients undergoing t-GES placement
determine the feasibility and patient tolerability of endoscopic placement of t-GES | 1 year
  Determine if placement of t-GES is feasible and if the patients tolerate the t-GES

CONTACTS AND LOCATIONS:
Overall Officials: John M Wo, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Hosptial, Indianapolis, Indiana, United States